CLINICAL TRIAL: NCT07114952
Title: The Effect of Alternate Nasal Breathing Exercise on Blood Pressure and Stress Levels in Individuals With Hypertension: A Randomized Controlled Experimental Study
Brief Title: The Effect of Alternate Nasal Breathing Exercise ın Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University (Other)
Collaborators: Cukurova University (Other)
Responsible Party: Principal Investigator, Leyla Senem Ün, Research assistant, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CU-SBF-LSU-01
Record Dates: First submitted 2025-07-29; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Hypertension (HTN)
Keywords: Hypertension; Breathing Exercises; Blood pressure; Stress; Nursing
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: "In this randomized controlled trial, participants were divided into two groups: an intervention group performing alternate nasal breathing exercises and a control group with no intervention. Outcomes were measured before and 4 weeks after the intervention period."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- alternative nasal breathing exercise intervention group (Experimental): The intervention group of 26 participants practiced an alternative nasal breathing exercise. This group practiced alternate nasal breathing exercise for 4 weeks.
  Interventions: Behavioral: alternative nasal breathing
- control group (No Intervention): The group consisted of 26 participants. No intervention was administered. Participants continued their usual care without any additional exercises or treatments during the study period.

INTERVENTIONS:
Behavioral: alternative nasal breathing — The alternate nasal breathing exercise involves breathing in and out through both nostrils in a certain pattern and for a certain period of time. For example, an individual who breathes in through the right nostril for 5 seconds with the left nostril closed, then closes the right nostril and exhales through the left nostril for 5 seconds. Then he/she inhales through the left nostril for 5 seconds and exhales through the right nostril. A total of 6 breaths are taken per minute. The application is applied for 5 minutes, the patient rests in a calm environment for two minutes and the application is performed for another 5 minutes. In order to increase the compliance of individuals with the application, a sample video was watched and application instructions were given by the researcher. The application was performed while the patients were in an upright sitting position.
  Arms: alternative nasal breathing exercise intervention group

SUMMARY:
This study is a randomized controlled experimental trial designed to examine the effect of alternative nasal breathing exercises on blood pressure and perceived stress levels in patients with hypertension. The study sample includes a total of 52 patients, with 26 in the intervention group and 26 in the control group.

DETAILED DESCRIPTION:
Aim: This study is being conducted as a randomized controlled experimental study to examine the effect of alternate nasal breathing exercises on blood pressure and stress levels in hypertensive patients.

Materials and Methods: The study sample consists of 52 patients (26 intervention and 26 control) from cardiology outpatient clinics. Ethics committee approval, institutional permissions, and verbal and written informed consent were obtained from the participants. Patients in the intervention group are instructed to perform alternate nasal breathing exercises for 10 minutes daily for four weeks, while the control group continues with routine treatment. Data collection tools include the Patient Introduction Form, Perceived Stress Scale, Life Findings Follow-up Form, and Blood Pressure Monitoring Forms. Planned statistical analyses include Independent Sample t-test, Paired Sample t-test, chi-square test, Mann-Whitney U test, and Wilcoxon test.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65,
* Literate,
* Diagnosed with hypertension at least 6 months ago,
* No change in hypertension medications in the last three months,
* Functionally capable of performing alternative nasal breathing exercises,
* Patients who volunteered to participate in the study were included.

Exclusion Criteria:

* Patients with psychiatric diagnoses,
* Patients with cognitive impairment,
* Patients practicing yoga or breathing exercises for hypertension,
* Patients with heart failure, cancer, kidney failure, or respiratory diseases were not included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure | Baseline and 4 weeks after intervention
  The blood pressure of the patients in the control group was measured twice, at the beginning of the study and 1 month later. In the measurement to be performed in the morning hours, the patients rested for 5 minutes in a calm environment before the measurement and then the measurement was made from the brachial artery in the arm. The same automatic sphygmomanometer was used for blood pressure measurement in all patients. " https://www.stridebp.org/bp-monitors/ " A blood pressure measuring device listed at

SECONDARY OUTCOMES:
Change in perceived stress scores | Baseline and 4 weeks after intervention
  The Perceived Stress Scale was used to assess perceived stress. The 10-question form was used in our study. The scale has a two-factor structure consisting of perceived inadequacy/self-efficacy and stress/distress. Responses are based on a five-point Likert scale, ranging from never (0) to very often (4), with reverse-scored items (4, 5, 7, 8). As the score from the scale increases, stress levels also increase.
Change in self-measured home blood pressure | Daily measurements during the 4-week intervention period
  Blood pressure measurements at home were taken using automatic blood pressure monitors. Patients were instructed on blood pressure measurement rules, such as taking measurements two hours after breakfast and after resting for five minutes, and were given a home blood pressure monitoring form to ensure follow-up. The form, which is intended for blood pressure monitoring, also ensures communication between the researcher and the patient.
  The four-week form includes patients' home blood pressure measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Adana City Training and Research Hospital, Cardiology Outpatient Clinic, Adana, Yüreğir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No